CLINICAL TRIAL: NCT05135442
Title: The Efficacy and Safety of Bortezomib as First-line Treatment for Acquired Thrombotic Thrombocytopenic Purpura
Brief Title: Efficacy and Safety of Bortezomib as First-line Treatment of Acquired TTP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FTTPB
Record Dates: First submitted 2021-11-06; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Thrombotic Thrombocytopenic Purpura, Acquired
Keywords: thrombotic thrombocytopenic purpura; bortezomib; plasma exchange
MeSH Terms: conditions — Thrombotic thrombocytopenic purpura, acquired; Purpura, Thrombotic Thrombocytopenic | interventions — Bortezomib; Plasma Exchange

STUDY DESIGN:
Intervention Model Description: Clinically diagnosed as TTP (thrombocytopenia + MAHA± clinical evidence of related organ damage), confirmed by ADAMTS13 activity level decreased significantly and/or positive antibody screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- bortezomib group (Experimental): On the basis of standard single membrane plasma exchange (2L/d) and hormone therapy (1mg/kg prednisone or equivalent methylprednisolone), bortezomib was given intravenous injection of 1.3mg/m2 d1, 4, 8, 11 (total 4 doses).
  Interventions: Drug: Bortezomib Injection

INTERVENTIONS:
Drug: Bortezomib Injection — Bortezomib should be administered immediately after each plasma exchange, and the interval between the next plasma exchange is> 24h. Plasma exchange continued until the patient's platelet count was >100×109/L for 2 consecutive days, and then changed to once every other day for a total of two times and then stopped.
  Other Names: plasma exchange; hormone therapy

SUMMARY:
To evaluate the efficacy and safety of bortezomib in the first-line treatment of patients with acquired TTP，we design this prospective, multi-center, single-arm interventional study.All enrolled TTP patients were given bortezomib 1.3 mg/m2 intravenous injection d1, 4, 8, on the basis of standard single membrane plasma exchange (2L/d) and hormone therapy (1mg/kg prednisone or equivalent methylprednisolone). 11 (4 doses in total). Bortezomib should be administered immediately after each plasma exchange, and the interval between the next plasma exchange is> 24h. Plasma exchange continued until the patient's platelet count was >100×109/L for 2 consecutive days, and then changed to once every other day for a total of two times and then stopped.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of bortezomib in the first-line treatment of patients with acquired TTP，we design this prospective, multi-center, single-arm interventional study.All enrolled TTP patients were given bortezomib 1.3 mg/m2 intravenous injection d1, 4, 8, on the basis of standard single membrane plasma exchange (2L/d) and hormone therapy (1mg/kg prednisone or equivalent methylprednisolone). 11 (4 doses in total). Bortezomib should be administered immediately after each plasma exchange, and the interval between the next plasma exchange is> 24h. Plasma exchange continued until the patient's platelet count was >100×109/L for 2 consecutive days, and then changed to once every other day for a total of two times and then stopped.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed as TTP (thrombocytopenia + MAHA± clinical evidence of related organ damage， a significant reduction in ADAMTS13 activity level and/or positive antibody screening）
* elder than 18 years old;
* informed consent is required;

Exclusion Criteria:

* Uncontrollable systemic infection;
* Known allergy to bortezomib;
* Expected survival time <1 week;
* Pregnant or lactating women (women of childbearing age have a positive pregnancy test at baseline or have not received a pregnancy test. Postmenopausal women must be at least 12 months after menopause);
* If the creatinine level is ≥200μmol/l (1.5mg/dl), the levels of transaminase and bilirubin are 2 times higher than the upper limit of normal (except due to the primary disease);
* Known congenital TTP or a clear family history of TTP;
* Other diseases that cause microangiopathic hemolysis and thrombocytopenia, such as DIC, APS, HUS, malignant hypertension, transplantation-related microangiopathy;
* active malignant tumors (except skin basal cell carcinoma or cervical carcinoma in situ) ( have not been treated or recurred within 5 years before signing the informed consent);
* peripheral neuropathy;
* Patients or family members cannot understand the conditions and goals of this study;
* The investigator believes that the patient should not participate in any other situations in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical remission and the number of plasma exchanges required | one month
  clinical remission means clinical symptom remission and/or adamts13 antibody negative，time to clinical remission means the days from first plasma exchange to clinical remission. the number of plasma exchanges required means the whole number of plasma exchanges in this course of TTP.

SECONDARY OUTCOMES:
Mortality rate | 6 months
  The ratio of the number of deaths to the total number of cases
ICU hospitalization time and total hospitalization time; | 6 months
  ICU hospitalization time means Duration of treatment in the ICU during the course of the disease(the number of days), total time in hospital(the number of days)

CONTACTS AND LOCATIONS:
Overall Officials: tienan zhu, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, (Select), China

REFERENCES:
- [Background] Scully M, Cataland S, Coppo P, de la Rubia J, Friedman KD, Kremer Hovinga J, Lammle B, Matsumoto M, Pavenski K, Sadler E, Sarode R, Wu H; International Working Group for Thrombotic Thrombocytopenic Purpura. Consensus on the standardization of terminology in thrombotic thrombocytopenic purpura and related thrombotic microangiopathies. J Thromb Haemost. 2017 Feb;15(2):312-322. doi: 10.1111/jth.13571. Epub 2017 Jan 30. PMID 27868334
- [Background] Patriquin CJ, Thomas MR, Dutt T, McGuckin S, Blombery PA, Cranfield T, Westwood JP, Scully M. Bortezomib in the treatment of refractory thrombotic thrombocytopenic purpura. Br J Haematol. 2016 Jun;173(5):779-85. doi: 10.1111/bjh.13993. Epub 2016 Mar 24. PMID 27009919
- [Background] Shortt J, Oh DH, Opat SS. ADAMTS13 antibody depletion by bortezomib in thrombotic thrombocytopenic purpura. N Engl J Med. 2013 Jan 3;368(1):90-2. doi: 10.1056/NEJMc1213206. No abstract available. PMID 23281998